CLINICAL TRIAL: NCT05542277
Title: A Pre-market, Multi-center, International, Double-blind, Randomized, Two-arms, Controlled, Prospective Clinical Investigation Assessing the Safety and Performance of a Medical Device (ClearPlasma™) for the Treatment of Patients Undergoing Coronary Artery Bypass or Valve Replacement
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: The study was stopped to evaluate the differences between the indications.
Sponsor: PlasFree Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: PLAS-01-2021
Record Dates: First submitted 2022-08-19; First posted 2022-09-15 (Actual); Last update posted 2025-06-15 (Actual); Status verified 2023-12

CONDITIONS: Bleeding; Bypass Complication; Valve Replacement
MeSH Terms: conditions — Hemorrhage

STUDY DESIGN:
Intervention Model Description: Multi-center, international, double-blind, randomized, controlled, prospective, clinical investigation, in which Patients undergoing Coronary Artery Bypass Grafting or valve replacement surgeries with a cardiopulmonary bypass, required plasma transfusion, will be randomized to receive a one-time infusion (up to 12 hours) of PDP (group A) or FFP (group B) with unlimited number of plasma units. The administration of plasma needs to be in line with the clinical practice and doctor decision. Furthermore, the main point is the patients with CABG/VRS that lost significant blood and need transfusion. Patients will be continuously monitored during transfusion and during stay in ICU. The assessment and additional test will be done at the admission to the ICU, 12 hours (±1) after procedure, 24 hours (±1) after procedure, 48 hours (±2) after procedure, at the discharge and 30±3 days after procedure.
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: After all applicable screening assessments have been performed, patients who have met all inclusion criteria and none of the exclusion criteria will be randomly allocated to one of the two treatment groups (with ratio 1:1) and will receive a unique computer-generated randomization number. Site stratified block randomization will be used during the study. Blocks length will have random length (e.g., 4, 6, 8). In order to reduce bias as much as possible, the trial will be double-blinded, keeping Sponsor, all patients and the Investigator blinded to the treatment. The randomization list will not be available to blinded personnel (such as Principal Investigator) involved in the conduct and evaluation of the trial until the trial database is locked.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- ClearPlasma (Experimental): Investigational Group (A): one-time infusion (up to 12 hours after surgery) of unlimited plasminogen depleted plasma PDP units generated by ClearPlasma™ device.
  Interventions: Device: ClearPlasma
- Control (Placebo Comparator): Control Group (B): one-time infusion (up to 12 hours) of unlimited regular plasma, Fresh frozen plasma (FFP) with mock ClearPlasma™ device.
  Interventions: Device: ClearPlasma

INTERVENTIONS:
Device: ClearPlasma — ClearPlasma ClearPlasma™ is an extra-corporeal plasma filtration device, designed to specifically extract plasminogen, a protein that drives fibrinolysis, from up to 250 mL of plasma. ClearPlasma™ is a non-pyrogenic, sterile, single-use medical device

SUMMARY:
Bleeding is a significant complication in cardiac surgery, with 10-15% of open cardiac surgery patients experiencing major intra- or post-operative bleeding. To address this unmet need, PLAS-FREE LTD has developed ClearPlasma™, a single-use, extracorporeal plasma filtration device which extracts plasminogen from plasma to reduce fibrinolysis. The resulting plasminogen-depleted plasma (PDP) is expected to reduce risk of fibrinolysis and bleeding in patients undergoing plasma transfusions.

DETAILED DESCRIPTION:
Bleeding is a significant complication in cardiac surgery, with 10-15% of open cardiac surgery patients experiencing major intra- or post-operative bleeding. Bleeding complications are associated with worse clinical outcomes, including a higher risk of infection, ischemic events attributable to hypo-perfusion (e.g., myocardial infarction, acute kidney injury), in-hospital mortality, and transfusion-related adverse events. Additionally, bleeding complications are an important driver of blood product utilization in cardiac surgery. Coagulopathy and bleeding after cardiac surgery are often a multifactorial problem, thus there is unmet need to find new technologies that can give better care to these bleeding patients. In 2016, it was estimated that one million people throughout the world undergo cardiac surgery each year. Most of these surgeries are Coronary artery bypass grafting and valves replacement. Coronary artery bypass grafting (CABG) is still the most commonly performed cardiac surgery procedure worldwide, representing annual volumes of approximately 200,000 isolated cases in the US and an average incidence rate of 62 per 100,000 inhabitants in western European countries. Aortic valve replacement is procedure that treat diseases affecting the aortic valve, one of four valves that control blood flow through the heart. In the United States, it is estimated that 2.5% of the general population, 8.5% of those 65-74 years of age and 13.2% of those ≥75 years of age have moderate to severe valvular diseases. These surgeries are commonly done in the western countries, however, the ability to halt the bleed remain challenge for most clinicians. Failed or delayed treatment of a massive bleeding can result in irreversible end-organ damage (e.g., renal failure), cardiovascular events (e.g., stroke, myocardial injury) or death, accompanied by significantly increased costs.

Fibrin clot breakdown is actively mediated by plasmin, a serine protease which cleaves fibrin. Administration of plasma depleted of plasminogen, the precursor of plasmin, may shift the balance towards coagulation.

PLAS-FREE LTD has developed ClearPlasma™, a single-use, extracorporeal plasma filtration device which extracts plasminogen from plasma to reduce fibrinolysis. The resulting plasminogen-depleted plasma (PDP) is expected to reduce risk of fibrinolysis and bleeding in patients undergoing plasma transfusions.

ELIGIBILITY:
Inclusion Criteria:

1. Patients aged ≥ 18 years
2. Patients undergoing isolated coronary artery bypass grafting or valve replacement surgeries with a cardiopulmonary bypass
3. Patients that need at least 2 units of plasma transfusion according to the physician's decision.
4. Patients understanding the nature of the study and providing their informed consent to participation;
5. Patients willing and able to attend the follow-up visits and procedures foreseen by study protocol.

   -

Exclusion Criteria:

1. Patients who underwent a plasma infusion in the 30 days before enrolment;
2. Patients in a life-threatening condition at the time of enrolment;
3. Patients who are hemodynamically unstable and required pressor administration at the time of enrolment (i.e. hypovolemic shock, cardiogenic shock);
4. Transfusion of cryoprecipitate during procedure.
5. Patients suffering from Hemophilia A or B;
6. Patients suffering from venous and arterial thromboembolic events within 3 months before the enrolment;
7. Patients with increased risk of blood clotting, according to Investigator's judgement;
8. Patients with fluid accumulation in the brain at the time of enrolment.
9. Patients with retinal thrombosis at the time of enrolment;
10. Patients with history of allergic reaction to plasma, polyethersyplone or polycarbonate;
11. Patients suffering from known IgA deficiency at the time of enrolment;
12. Patients identified by the Investigator to have any underlying medical conditions that may preclude conduct of study procedure (i.e. making the administration of study treatment hazardous) or obscure the interpretation of safety objectives;
13. Patients who are participating or have participated in other clinical studies within the 30 days before the study enrolment.
14. Women who are pregnant or breast-feeding or who wish to become pregnant during the period of the clinical investigation and for 3 months later;
15. Female Patients of childbearing age (less than 12 months after the last menstrual cycle) who do not use adequate contraception*.

Methods at low risk of contraceptive failure (less than 1% per year) when used consistently, including: combined (estrogen and progestogen containing) hormonal contraception associated with inhibition of ovulation (oral, intravaginal, transdermal), progestogen-only hormonal contraception associated with inhibition of ovulation (oral, injectable, implantable), some intra-uterine devices.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2022-11-08 (Actual); Primary Completion 2025-03-09 (Actual); Study Completion 2025-03-09 (Actual)

PRIMARY OUTCOMES:
ClearPlasma efficacy | 30 days
  Post-operative blood loss (mL) within 24 hours after surgery, defined as total output of mediastinal and pleural chest tubes. [time frame: up to 24 hours after procedure]

SECONDARY OUTCOMES:
Transfusion- related SAE | 30 days
  Comparison of the number of transfusion- related SAEs between the groups. [time frame: discharge]obtained through filtration with ClearPlasma™ in patients after coronary artery bypass grafting or valve replacement surgery and to compare it to the same procedure carried out using FFP units.
Hemoglobin levels | 30 days
  Comparison of hemoglobin levels drop between the groups [time frame: measured at patient's departure from the operating room/admitting to the ICU and compared to the lowest hemoglobin value until discharge]
Post-operative blood loss | 30 days
  Post-operative blood loss (mL) within 12 hours after surgery, defined as total output of mediastinal and pleural chest tubes. [time frame: up to 12 hours after procedure]
Total blood loss | 30 days
  Total blood loss, defined as total output of chest tubes from insertion till removal [time frame: drain removal]
ClearPlasma | 30 days
  Ratio of bleeding events between the groups [time frame: discharge]
bleeding events- | 30 days
  Ratio of bleeding events requiring re-intervention up to discharge [time frame: discharge]
major bleeding | 30 days
  Ratio of major bleeding defined as blood loss greater than >1000 mL in first 12 h and/or need for surgical revision owing to bleeding; [time frame: discharge]
Mortality | 30 days
  All-cause mortality[time frame: 30 days]
In- hospital mortality | 30 days
  In- hospital mortality [time frame: discharge]
Number of blood units transfused | 30 days
  The number of units of allogeneic blood products transfused until discharge [time frame: discharge]:
  1. Red blood cells (RBC) units transfused;
  2. Plasma (PDP/FFP) units transfused;
  3. Platelet concentrates units transfused
Length of stay in the ICU | 30 days
  Length of stay in the ICU [Time Frame: discharge]
Hospitalization Duration | 30 days
  Total length of hospitalization [Time Frame: discharge]
Incidence of ischemic outcomes | 30 days
  Comparison of the incidence of ischemic outcomes defined as a composite of stroke, transient ischemic attack, acute myocardial infarction, PE and/or acute renal failure [time frame: discharge] Study Groups

CONTACTS AND LOCATIONS:
Overall Officials: Zeev Dvashi, Ph.D, Study Director — Plas-Free LTD
Locations (8):
- Czechia (3):
  - Charles University Teaching Hospital, Hradec Králové
  - University Hospital Olomouc, Olomouc
  - University Hospital Ostrava, Ostrava
- Israel (3):
  - Wolfson Medical center, Holon
  - Rabin Medical Center - Beilinson, Petah Tikva
  - Sheba Medical Center, Ramat Gan
- Poland (2):
  - Szpital Kliniczny im. Heliodora Święcickiego Uniwersytetu Medycznego w Poznaniu, Poznan
  - Narodowy Instytut Kardiologii Stefana kardynała Wyszyńskiego Państwowy Instytut Badawczy, Warsaw

IPD SHARING:
Plan to Share IPD: Yes
all data will be published in peer review article
Supporting Information: Study Protocol
Time Frame: 1 year after the study will end
URL: http://www.Plas-free.com